CLINICAL TRIAL: NCT04834791
Title: Letrozole Versus Gonadotropins for Ovulation Induction in Clomiphene Citrate Resistance: A Randomized Controlled Study
Brief Title: Letrozole Versus Gonadotropins in Clomiphene Citrate Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Clomiphene Citrate Resistance; Ovulation Induction; Letrozole; Gonadotropins
MeSH Terms: interventions — Letrozole; Gonadotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole (Experimental): These patients were treated with letrozole (Femara®, Novartis New York, NY, USA) in a dose 2.5 mg (one tablet daily) orally began on the 3rd day to the 7th day of the cycle. If ovulation is not achieved dose is increased by 2.5 mg in next cycle till 3 cycles.
  Interventions: Drug: Letrozole 2.5mg
- Gonadotropins (Active Comparator): These patients were given urofollitropin (fostimon ®, IBSA, Lugano, Switzerland) in a dose of 75 IU/mL I.M from day 3rd to day 7th of the cycle beginning by one ampoule per day and the dose had been modulated according to response.
  Interventions: Drug: Gonadotropin

INTERVENTIONS:
Drug: Letrozole 2.5mg — These patients were treated with letrozole (Femara®, Novartis New York, NY, USA) in a dose 2.5 mg (one tablet daily) orally began on the 3rd day to the 7th day of the cycle. If ovulation is not achieved dose is increased by 2.5 mg in next cycle till 3 cycles
  Arms: Letrozole
Drug: Gonadotropin — These patients were given urofollitropin (fostimon ®, IBSA, Lugano, Switzerland) in a dose of 75 IU/mL I.M from day 3rd to day 7th of the cycle beginning by one ampoule per day and the dose had been modulated according to response.
  Arms: Gonadotropins

SUMMARY:
Clomiphene citrate resistance (CCR) occur in 15-40% in women with PCOS. Several studies have shown that letrozole is superior to CC regarding side effects, ovulation, and pregnancy rates. Letrozole or gonadotropins use for ovulation induction in CCR is not well established which is superior and most safe.

DETAILED DESCRIPTION:
This study included 70 patients enrolled according inclusion and exclusion criteria. The inclusion criteria were (a) Infertility lasting one year or more in presence of regular intercourse, (b) Patients' age between 20-35years (c) Normal semen analysis according to WHO 2010 (d) Patent fallopian tubes (e) Normal prolactin and TSH. (e) Anovulatory cycles confirmed by mid-luteal progesterone ≤ 3 ng/ml and (f) Clomiphene citrate resistance for 3 cycles of 150mg. Exclusion Criteria were (a) Any hormonal disturbances eg. hyperprolactinemia, (b) Immunological causes of infertility, (c) Coital errors, (d) Metabolic disorders and (e) Poor patient compliance.

Sample size calculation: The minimum sample size calculated using Epi info program version 7 for unmatched case control study; 80% power and 95% Confidence interval was 22 for each group. For better accuracy and validity of results the sample size was increased by 10%=3 in each group. The total number of cases was 50 and 25 for each group.

Randomization and allocation: It was a prospective quesi-randomization. Based on the attendance order, patients with odd numbers were considered group I (Letrozole group) and those with even numbers were considered group II (Gonadotropin group). Allocation was equal 1:1.

Intervention:

Group I (Letrozole Group n=25): These patients were treated with letrozole (Femara®, Novartis New York, NY, USA) in a dose 2.5 mg (one tablet daily) orally began on the 3rd day to the 7th day of the cycle. If ovulation is not achieved dose is increased by 2.5 mg in next cycle till 3 cycles. If hyperstimulation occurred, the cycle was cancelled and the patients were excluded from the study.

Group II (Gonadotropin Group n=25) These patients were given urofollitropin (fostimon ®, IBSA, Lugano, Switzerland) in a dose of 75 IU/mL I.M from day 3rd to day 7th of the cycle beginning by one ampoule per day and the dose had been modulated according to response. If hyperstimulation occurred, the cycle was cancelled and the patients were excluded from the study.

Methods:

Proper history taking including age, gravidity, parity, infertility duration, history of laparoscopic surgery, previous induction of ovulation in the last 6 months. Examination was done to assess weight, height (BMI), signs of androgen excess, thyroid gland and breast examination.

Serum FSH, LH, testosterone level, prolactin level and thyroid stimulating hormone on day 3 of spontaneous menstrual cycle were done. Serum Progesterone (P4) was done on day 22 (midluteal) to confirm ovulation if ≥ 10ng/ml.

Basal transvaginal U/S on day3 of the cycle to detect criteria of PCOS and count number of antral follicles in both ovaries and to exclude of any basal ovarian cyst. Transvaginal ultrasound was also used to follow follicular growth and endometrial thickness starting on day 8 and then every other day till assuming good ovulatory response when one or more follicles is ≥ 18mm and endometrial thickness ≥ 6mm.

Human Chorionic Gonadotropin (choriomon®, IBSA, Lugano, Switzerland) 10.000IU/I.M was administered when good ovulatory response was assumed. The intercourse was advised on the day of HCG injection and every other day for 4 days after injection HCG.

Number and size of Dominant follicles, endometrial thickness were recorded. Clinical pregnancy was detected by serum pregnancy test and by presence of intrauterine gestational sac with fetal pulsation.

Outcome measures: Primary outcomes was ovulation rate. Secondary outcomes were pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Infertility lasting one year or more in presence of regular intercourse,
* Patients' age between 20-35years
* Normal semen analysis according to WHO 2010
* Patent fallopian tubes (e) Normal prolactin and TSH.
* Anovulatory cycles confirmed by mid-luteal progesterone ≤ 3 ng/ml and
* Clomiphene citrate resistance for 3 cycles of 150mg.

Exclusion Criteria:

* Any hormonal disturbances eg. hyperprolactinemia,
* Immunological causes of infertility,
* Coital errors,
* Metabolic disorders and
* Poor patient compliance.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 6 months
  Number of mature follicles in each ovary>18mm

SECONDARY OUTCOMES:
Pregnancy rate | 6 months
  Number of pregnant women evidenced by serum HCG and gestational sac inside the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Dawood, MD, Principal Investigator — Assistant professor
Locations (1):
- Ayman Shehata Dawood, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
on request
Supporting Information: Study Protocol
Time Frame: 3 months